CLINICAL TRIAL: NCT06372093
Title: Evaluation of Bilirubin Measurements in Newborns From Smartphone Digital Images in a Population in Botswana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Picterus AS (Industry)
Collaborators: University of Copenhagen (Other); University of Botswana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PMH 2/11AII
Record Dates: First submitted 2024-01-22; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Jaundice, Neonatal
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enable reliable measurement of bilirubin levels in the blood of newborns (Experimental): to enable reliable measurement of bilirubin levels in the blood of newborns independent of skin color
  Interventions: Device: Picterus Jaundice Pro

INTERVENTIONS:
Device: Picterus Jaundice Pro — Picterus Jaundice Pro is a smartphone based screening tool for neonatal jaundice that takes images of the skin of the newborn chest where the Picterus Calibration Card is placed.
  Other Names: Picterus JP

SUMMARY:
The general objective of this study is to evaluate the accuracy of a novel smartphone application for jaundice screening (Picterus Jaundice Pro) in a population with high melanin content in the skin.

The specific objectives for this study are:

i. To assess the correlation between bilirubin level measurements obtained by Picterus Jaundice Pro with Total Serum Bilirubin (TSB), and TcB, in newborns with high melanin content in the skin.

ii. To determine the accuracy of Picterus Jaundice Pro in newborns with high melanin content in the skin.

DETAILED DESCRIPTION:
The goal for this project is to demonstrate that the Picterus Jaundice Pro screening method can be used to identify children with severe neonatal jaundice independent of skin color. Thus, providing a cheaper, patient-friendly, and more readily available method of neonatal jaundice detection. The long-term goal is that with the implementation of the app, the identification of newborns with severe jaundice will be improved and, thus, referred at an earlier stage for diagnostics and treatment.

The study will be a cross-sectional study with quantitative methods of data collection.

The study population will comprise 150 newborns from the Neonatal Unit and the maternity ward at Princess Marina Hospital.

Parents to newborns with and without signs of jaundice will be asked to participate.

Following informed consent, background data such as birth weight, age on examination, gestational age, and type of feeding will be obtained. Gestational age will be based on ultrasound determination and the last normal menstruation period (LNMP). The skin type of the infant will be classified according to the newborn Neomar's scale score.

Transcutaneous bilirubin measurements will be performed over the sternum of the infant. A Dräger Jaundice Meter JM-105 will be used in this study. Skin reflectance will be measured using a portable Konica Minolta spectrophotometer CM-700d.

A validated smartphone with Picterus Jaundice Pro will be used to collect digital images of skin of the infant chest together with the Picterus calibration card. After all the images are obtained, a unique ID will be displayed on the smartphone. This ID will be recorded on the case report forms and later used to pair clinical data and digital images.

A blood sample to determine TSB will be obtained within 60 minutes of obtaining the images and processed at the Department of clinical biochemistry in the hospital laboratory.

After completion of the study the bilirubin measurement from Picterus Jaundice Pro will be determined and compared to the TSB and TCB measurements using the Pearson correlation coefficient. Sub-analysis for the different skin colors will be performed. Systematic over- or under-estimation of bilirubin levels will be evaluated using Bland-Altman plots. Sensitivity and specificity analysis will be calculated for different cut-off values (ROC analysis).

ELIGIBILITY:
Inclusion Criteria:

* Gestational age > 37 weeks
* Birth weight > 2000 g and < 4500 g
* Age 1-14 days
* Infants requiring a blood sample for clinically suspected jaundice/screening

Exclusion Criteria:

* Infants transferred to the pediatric ward for advanced treatment.
* Infants with a skin rash or other disease that affects the skin where measurements are performed.
* Infants that receive or have received phototherapy in the last 24 hours.
* Infants with an inborn disease.

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Enable high qualitative estimation of bilirubin levels in the blood of newborns in a population in Botswana using Picterus JP. | 1 year
  Evaluate of smartphone-based screening tool (Picterus JP) for neonatal jaundice in newborns with high melanin content.

SECONDARY OUTCOMES:
Correlation of bilirubin levels obtained by Picterus JP with Tsb and TcB | 1-2 hours
  Correlate estimates of bilirubin levels obtained by Picterus JP with TSB and TcB in newborns with high melanin content in the skin.
Sensitivity and specificity of Picterus JP to detect jaundice in newborns with high melanin content in the skin | 1 year
  Determine the sensitivity and specificity of Picterus JP to screen for jaundice in newborns with high melanin content in the skin

CONTACTS AND LOCATIONS:
Overall Officials: Julie Zimmer, Principal Investigator — University of Copenhague; Britt Nakstad, MD, PhD, MSC, Study Director — Princess Marina Hospital
Locations (1):
- Princess Marina Hospital, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: No